CLINICAL TRIAL: NCT05834309
Title: Effectiveness of a Multicomponent Exercise Program on Health Status and Health-related Quality of Life in Patients With Severe Mental Illness: Study Protocol for a Randomized Controlled Trial.
Brief Title: Exercise Effects on Health Status in Patients With Severe Mental Illness
Acronym: SMI01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: Fundacion Miguel Servet (Other); Complejo Hospitalario de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UPNavarra
Record Dates: First submitted 2023-03-07; First posted 2023-04-28 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Exercise; Metabolic Syndrome; Mental Disorders, Severe; Severe Mental Disorder; Mental Deterioration; Physical Inactivity; Physical Disability; Health-Related Behavior
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome; Mental Disorders; Cognitive Dysfunction; Sedentary Behavior; Health Behavior | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in this group will receive clinical usual care.
- Exercise training group (Experimental): An individualized multicomponent exercise program including resistance, aerobic, balance and flexibility exercises.The duration of the sessions will be 45 minutes, and the duration of the whole program will be 6 weeks, equivalent to 12 sessions.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — The intervention protocol consists of a 10-minute warm-up doing joint mobility exercises and adaptation exercises to the core exercises of the training session. The exercises will be performed at low intensity in the warm-up. During the main part of the training session, exercises will be performed on a stationary bike at a higher intensity than in the warm-up and strengthening exercises using weights and body weight exercises such as jumping jacks and squats will also be performed. All movements will be performed at 100% of the maximum speed reached in the propulsive phase (understood as executing the movement as fast as possible according to your muscular and functional capacity). The rests between sets will be between 1 and 2 minutes. At the end of the session, there will be a 5-minute return to calm by stretching.
  Arms: Exercise training group

SUMMARY:
People with severe mental disorders have a mortality rate 2 to 3 times higher than that of the general population, largely due to the presence of comorbidities, with a predominance of cardiovascular disease. This population has a higher risk of developing metabolic syndrome compared to the healthy population. Several factors are involved. The usual pharmacological treatment in people with severe mental disorder is a risk factor for the development of metabolic syndrome and deterioration of physical condition. This is generally compounded by poor health care, high-calorie diets, a sedentary lifestyle, difficulties in coping with life situations that generate emotional states (anxiety and/or depression) that result in unhealthy lifestyle habits related to food, activity, interpersonal relationships, sleep, consumption habits (tobacco, alcohol and drugs) and other environmental factors. Physical exercise has been proposed as one of the most effective treatments to reverse the negative consequences of low levels of physical activity in this population. However, the mechanism of action of exercise on health status and the optimal "dose" and intensity of exercise to achieve the greatest number of benefits with respect to cardiometabolic health in patients with severe mental disorder are unknown.The study will be carried out at the Mental Health Rehabilitation Unit of Navarra, a center under the Mental Health Management of Osasunbidea, where people between 18 and 65 years of age with a diagnosis of severe mental illness in a situation of clinical stability receive treatment.The sample will be composed of 100 participants from consecutive admissions to the Rehabilitation Unit. The subjects will be randomized into 2 groups; a control group that will receive the usual specialized care and an intervention group, which in addition to receiving the usual rehabilitation treatment, will undergo a 6-week multicomponent physical exercise program performed 2 days per week. The effects of exercise on the inflammatory profile, metabolic parameters, physical condition, cognitive function, vascular function, muscle strength, health-related quality of life, lifestyle habits (diet, activation, sleep, substance use) and mood will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* resident in Navarra
* diagnosis of severe mental disorder (DSM 5: Schizophrenia 295.90, Tr. Schizoaffective Disorder 295.70, Schizotypal Personality Disorder 301.22, Schizoid Personality Disorder 301.20, Schizophreniform Personality Disorder 295.40, Psychotic Disorder with Delusional Ideas 295.40, Psychotic Disorder with Delusional Ideas 295.40. Schizophreniform 295.40, Psychotic disorder with delusions 293.81, Psychotic disorder with hallucinations 293.82, Major depressive disorder 296.33, Bipolar disorder type I 296.44, Bipolar disorder type II 296.89, Obsessive Compulsive Disorder 300.
* primary nursing diagnosis NANDA and Virginia Henderson NOC 0099 Ineffective Health Maintenance
* at least one of the secondary nursing diagnoses 001 Nutritional Imbalance due to Excess, 003 Risk of Nutritional Imbalance due to Excess, 00096 Sleep Deprivation, 00146 Anxiety or 00168 Sedentary
* willing to voluntarily participate in the randomly assigned intervention, after signing the informed consent form.

Exclusion Criteria:

* acute illness that does not allow physical exercise sessions or assessments during the study
* medical contraindication that prevents physical exercise
* treatment with Interleukin-6 receptor antagonists (tocilizumab) during the last month due to drug interference with adaptations to cardiopulmonary exercise
* refusal to sign the informed consent form by the study subject
* impossibility of follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2025-05-05 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of metabolic syndrome | 14 weeks
  Any 3 of the 5 features: Waist circumference (> 102 cm men/ > 88 cm women),Elevated triglycerides (> 150 mg/dl), reduced HDL cholesterol (< 40 mg/dl men/ < 50 mg/dl women), elevated blood pressure(> 130 mmHg Systolic blood pressure or > 85 mmHg Diastolic blood pressure), and elevated fasting glucose (> 100 mg/dl) glucose.

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 14 weeks
  Physical activity questionnaire. LOW If not moderate or vigorous. MODERATE: 3 or more days of vigorous-intensity activity of at least 20 minutes per day OR b) 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day OR c) 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum T=total physical activity of at least 600 Metabolic equivalent of task (MET)-minutes/week. HIGH a) Vigorous-intensity activity on at least 3 days (20min minimum, achieving a minimum Total physical activity of at least 1500 MET-minutes/week or 7 or more days of any combination of walking, moderate-intensity or vigorous-intensity activities achieving a minimum Total physical activity of at least 3000 MET-minutes/week.
Muscle strength | 14 weeks
  Maximal dynamic strength (one-maximum muscle strength) was measured for four exercises (knee extension, leg press, row and bench press) using a Smart Strength machine (eGym GmbH, München, Germany). Results were expressed in kilograms.
European Quality of Life-5 Dimensions (EuroQol-5D) | 14 weeks
  Health related quality of life.The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The worse score is 0 and the best score is 100.
Physical condition | 14 weeks
  Graded exercise tests will be performed on a bicycle ergometer (Lode B.V., Groningen, The Netherlands) to determine the maximal oxygen uptake (VO2max), measured by ml/kg/min.
Beck questionnaire | 14 weeks
  Depression. The minimum value is 0 points and the maximum value is 63 points. Higher scores mean a worse outcome.
State Strait Anxiety Inventory (STAI) | 14 weeks
  Anxiety. The minimum score is 0 and the maximum score is 120. Higher scores means a worse outcome.
Positive And Negative Syndrome Scale (PANSS) | 14 weeks
  Positive and negative symptoms. Positive scale (minimum score is 7 and maximum score is 49), negative scale (minimum scale is 7 and maximum score is 49) and general psychopathology scale (minimum score is 16 and maximum score is 112 points). Higher scores means a worse outcome.
Screen for Cognitive Impairment in Psychiatry (SCIP) | 14 weeks
  Cognitive function. Memory, attention, executive function and processing speed.
Adverse events related to medication | 14 weeks
  Neurological side effects related to the medication assessed by the Side Effect Rating Scale.
Muscle mass | 14 weeks
  Muscle thickness by ultrasound examination
Densitometry | 14 weeks
  Body composition
Medication | 14 weeks
  Pharmacologic/antipsichotic treatment (i.e., pills consumption) associated with the disorder obtained by the medical history.
Blood pressure | 14 weeks
  Blood pressure will be assessed using a Vasera 2000 device (Fukuda Denshi, Japan).
Oviedo questionnaire | 14 weeks
  Sleep quality.The insomnia subscale ranges from 9 to 45, where a higher scores means increased severity of insomnia.
Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) | 14 weeks
  Health related quality of life.The SQLS-R4 is a self-report measure comprising 33 items from which two domains of quality of life, psychosocial feelings (22 items) and cognition and vitality (11 items) are derived. The items are scored on a 5-point frequency-response Likert scale (''never'', ''rarely'', ''sometimes'', ''often'', ''always''). A total score of both domains can also be calculated and individual domain and total scores are standardized by scoring algorithm to a 0 - 100 scale. Higher SQLS-R4 scores indicate comparatively lower quality of life.
The Matrics Consensus Cognitive Battery | At baseline
  Cognitive function.The MATRICS Consensus Cognitive Battery should be used as the standard battery for all clinical trials of potential cognition-enhancing agents for schizophrenia.
  * The battery should always be administered in its entirety in clinical trials (64 minutes).
  * An overall cognitive composite score consisting of equal weighting of the 7 domain scores is the primary cognitive endpoint for agents believed to enhance cognition broadly.
  * Alternatively, a small subset of domains may be combined as the primary cognitive endpoint for agents believed to enhance cognition selectively (e.g., the learning and memory domains).
Medical history of substance abuse | 14 weeks
  Alcohol consumption, use of drugs and other substances.
Vascular stiffness | 14 weeks
  Cardio-ankle vascular index (CAVI) will be estimated by brachial-ankle oscillometry using a Vasera 2000 device (Fukuda Denshi, Japan) as marker of vascular stiffness.
Vascular stiffness | 14 weeks
  Pulse wave velocity (PWV) will be estimated by brachial-ankle oscillometry using a Vasera 2000 device (Fukuda Denshi, Japan).

CONTACTS AND LOCATIONS:
Overall Officials: Ana Urteaga, Principal Investigator — Complejo Hospitalario de Navarra
Locations (2):
- Spain (2):
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Fundacion Miguel Servet, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Undecided